CLINICAL TRIAL: NCT04313894
Title: THE EFFECTIVENESS of WHARTON JELLY ORIGINATED MESENCHIAL STEM CELL in TREATMENT of KNEE OSTEOARTHRITIS
Brief Title: WHARTON JELLY ORIGINATED MESENCHIAL STEM CELL in GONARTHROSIS
Acronym: WHAMKO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, İbrahim Karaman, TC Erciyes University - Scientific Researches Projects Support, TC Erciyes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/397
Record Dates: First submitted 2019-02-09; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Stem Cell; Gonarthrosis
Keywords: Gonarthrosis; Degenerative Arthritis Treatment; Stem Cell Therapia
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stem Cell Therapia Group (Experimental): A total of 11 patients with Kellgren-Lawrence grade II-III knee OA who were admitted to the outpatient clinic with knee pain and who had received conservative treatment for a period of 6 months and who had not benefited from it will be taken. Patients will be evaluated 7 (V1-7) during the study period. Patients who comply with the study criteria will be included in the study. The clinical, immunological and radiological efficacy of the treatment and clinical improvement will be evaluated in all follow-up patients at the beginning and at the beginning of the treatment.
  Interventions: Biological: Wharton Jelly Originated Mesencimal Stem Cell

INTERVENTIONS:
Biological: Wharton Jelly Originated Mesencimal Stem Cell — In this study, the patient who has no systemic disease from Erciyes University, Obstetrics and Gynecology Department will be taken to the cord transport solution which will be medical waste after delivery. Samples for transport bacteriological tests from the transport solution to the laboratory shall be separated. They will be processed in a number of ways. The cells obtained will be administered intraarticularly at a dose of 1 x 100.000.000.

SUMMARY:
Osteoarthritis (OA) is a progressive disease characterized by degeneration of the joint cartilage, which is involved in the immune system leading to proinflammatory cytokine and metalloproteinase release. Knee osteoarthritis is the most common form. The healing is very slow and the damage is not fully recovered, so the degeneration process continues and no treatment modalities completely remove this process. Various methods are used in the treatment of OA and total joint replacement is performed in the patients with OA recently.

Ten patients with Kellgren-Lawrence grade II-III knee OA who had been applied for knee pain and received conservative treatment for 6 months and had no benefit will be taken to study. Patients will be assessed 7 (V1-7) times during the study. Clinical, immunologic and radiological treatment effectiveness and clinical improvement will be evaluated at the beginning of the treatment and in all follow-up patients participating in the study.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a progressive disease characterized by degeneration of the articular cartilage, caused with the release of proinflammatory cytokines and metalloproteinases. Knee osteoarthritis is the most common form. OA accounts for about 2% of public health problems and leads to a reduction in production, resulting in indirect costs. Regardless of the etiology (age, trauma, overuse, autoimmune arthritis, infection, etc.), the recovery is very slow, the damage is not fully recovered, and the result is secondary fibrosis healing. Therefore, the degeneration process continues and no treatment modality does not completely eliminate this process. Various methods are used in the treatment of OA. The most commonly used of these methods are the physical and educational therapy offered by the American Society of Orthopedic Surgeons (AAOS), symptomatic treatment with acetaminophen and non-steroidal anti-inflammatory drugs, and steroid injection. In patients with end-stage OA who do not benefit from these treatment methods, total joint replacement is performed. Mesenchymal stem cells are multiple potent progenitor cells. In recent years, there have been promising developments in the treatment of patients who cannot be cured by stem cell therapy. Mesenchymal stem cells have been used in clinical and experimental animal studies due to their immunosuppressive effects, limited immunogenetic effects, their ability to be produced in culture and their multilevel structure. At the same time, studies have shown that mesenchymal stem cells have potential to differentiate into osteocytes, chondrocytes, muscle cells and nerve cells. Because of these features, mesenchymal stem cells have been used clinically for OA treatment. In addition, studies have shown that mesenchymal stem cells can be obtained from bone marrow, periosteum, trabecular bone, fat tissue, synovia, muscle tissue, milk tooth, umbilical cord and Wharton gel. Wharton gel is a mucous connective tissue in the umbilical cord and consists of myofibroblast-like stromal cells, collagen fibers, proteoglycans and hyaluronic acid. Because of these properties, it can be used as a source of stem cells.

dipocytokines are cytokines secreted from adipose tissue and act as intercellular signal proteins. These cytokines include adipose tissue and cells nutrient uptake, regulation of energy balance, insulin activation, lipid and glucose metabolism, angiogenesis, regulation of blood pressure, coagulation, immunostimulation, pro-inflammatory and anti-inflammatory effects.

Stem cell applications are now widely used in different tissues. In the recovery of chondral damage; Since cells have little capacity for regeneration and proliferation, stem cell derived differentiation is needed. In this study, it will be tried to show that chondral damage can be treated with wharton gel-derived stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Kellgren-Lawrence Grade II-III OA
* Between 60- 65 years old
* Those with chronic knee pain not undergoing 6 months of conservative treatment
* Body Mass Index: 25-30 kg / m2
* Patients who understand the content of the study
* Patients with written consent form

Exclusion Criteria:

* Patients with Diabetes Mellitus
* Patients with septic table
* Patients with bleeding diathesis
* Patients with HIV and Hepatitis
* Body Mass Index greater than 30 kg / m2 and lower than 25 kg / m2
* Those with congenital axis disorder
* Those with malignancy
* Immunosuppressive
* Lumbar pathological findings

Ages: 60 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changing of Pain after Wharton Jelly Originated Mesenchial Stem Cell İnjection for one year | Before injection and 15 Day - 30 Day - 45 Day - 3 months - 6 Months - 12 Months after injection
  Pain Evaluation With Visual Analog Scale (min : 0 - max: 10)
Changing of functional knee score after Wharton Jelly Originated Mesenchial Stem Cell İnjection for one year | Before injection and 15 Day - 30 Day - 45 Day - 3 months - 6 Months - 12 Months after injection
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).
Changing of life Quality after Wharton Jelly Originated Mesenchial Stem Cell İnjection for one year | Before injection and 15 Day - 30 Day - 45 Day - 3 months - 6 Months - 12 Months after injection
  Short Form 36 (min :0 - max :100)
Radiological Changings according to Kellgren-Lawrence classification systemafter Wharton Jelly Originated Mesenchial Stem Cell İnjection for one year | Before injection and 12 Months after injection
  Direct Graphy Kellgren-Lawrence classification (0-4) - (0 : Better)
Chondral and subchondral Changings after Wharton Jelly Originated Mesenchial Stem Cell İnjection for one year | Before injection and 12 Months after injection
  Magnetic Resosonans Imaging T2 mapping (msn): If an area have a value above 50/msn that will named as inflamated cartilage. This area's size and mean speed will be evaluated.
Changing of Leptin levels in sinovial fluid after Wharton Jelly Originated Mesenchial Stem Cell İnjection for one year | Before injection and 15 Day - 30 Day - 45 Day - 3 months - 6 Months - 12 Months after injection
  Leptin levels in sinovial fluid (elisa)
Changing of adiponectin levels in sinovial fluid after Wharton Jelly Originated Mesenchial Stem Cell İnjection for one year | Before injection and 15 Day - 30 Day - 45 Day - 3 months - 6 Months - 12 Months after injection
  Adiponectin levels in sinovial fluid (elisa)
Changing of tumor necrosing factor-α levels in sinovial fluid after Wharton Jelly Originated Mesenchial Stem Cell İnjection for one year | Before injection and 15 Day - 30 Day - 45 Day - 3 months - 6 Months - 12 Months after injection
  tumor necrosing factor-α levels in sinovial fluid (elisa)
Changing of resistin levels in sinovial fluid after Wharton Jelly Originated Mesenchial Stem Cell İnjection for one year | Before injection and 15 Day - 30 Day - 45 Day - 3 months - 6 Months - 12 Months after injection
  Resistin levels in sinovial fluid (elisa)
Changing of interleukin-6 levels in sinovial fluid after Wharton Jelly Originated Mesenchial Stem Cell İnjection for one year | Before injection and 15 Day - 30 Day - 45 Day - 3 months - 6 Months - 12 Months after injection
  interleukin-6 levels in sinovial fluid (elisa)
Changing of interleukin-1β levels in sinovial fluid after Wharton Jelly Originated Mesenchial Stem Cell İnjection for one year | Before injection and 15 Day - 30 Day - 45 Day - 3 months - 6 Months - 12 Months after injection
  interleukin-1β levels in sinovial fluid

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim Karaman, Asc.Prof, Study Director — TC Erciyes University
Locations (1):
- Erciyes University Faculty of Medicine, Melikgazi, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided